CLINICAL TRIAL: NCT06356480
Title: RANDOMIZED CONTROL TRIAL TO COMPARE 1% ACETIC ACID DRESSING VS SALINE DRESSING TO SEE EARLY WOUND HEALING IN DIABETIC WOUNDS.
Brief Title: 1% Acetic Acid vs Normal Saline Dressing inManagement of Diabetic Foot
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Muhammad Naeem (Other)
Responsible Party: Sponsor-Investigator, Dr. Muhammad Naeem, Head of the department of surgery, Pak Emirates Military Hospital
Organization: Pak Emirates Military Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 266
Record Dates: First submitted 2024-03-22; First posted 2024-04-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Granulation of Chronic Diabetic Wounds; Diabetic Wounds
Keywords: Diabetic wounds, 1% acetic acid, epithelialization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1% acetic acid dressing in chronic diabetic wounds (Experimental): 1% Acetic acid dressing in chronic diabetic wounds twice daily along with oral antibiotics to see the early epithelialization of the wounds
  Interventions: Biological: 1% Acetic acid dressing
- Normal saline soaked dressing in chronic diabetic wounds (No Intervention): Normal Saline soaked dressing in chronic diabetic wounds along with antibiotics to see early epithelialization over diabetic wounds

INTERVENTIONS:
Biological: 1% Acetic acid dressing — 1% acetic acid dressing in chronic diabetic foot and wounds to see early epithelialization and later on graft application.
  Arms: 1% acetic acid dressing in chronic diabetic wounds

SUMMARY:
Chronic diabetic wounds are those wounds that are persistent and do not respond to any sort of treatment. The concept of using topical antiseptics on open wounds is to prevent and treat infections. They also help to shorten the time taken to heal the wounds. The use of topical agents on wounds to prevent infection is a minimal ability to develop resistance to the microorganisms. Pseudomonas aeruginosa is a Gram-negative opportunistic pathogen with innate resistance to many antibiotics. In places that are economically backward, these problems get compounded by the inability of patients to afford newer expensive drugs. Topically applied dilute acetic acid, which is cheap and easily available, has been found to be effective in such chronic diabetic wounds

DETAILED DESCRIPTION:
Chronic diabetic wounds are those wounds that are persistent and do not respond to any sort of treatment. The concept of using topical antiseptics on open wounds is to prevent and treat infections. They also help to shorten the time taken to heal the wounds. The use of topical agents on wounds to prevent infection is a minimal ability to develop resistance to the microorganisms. Pseudomonas aeruginosa is a Gram-negative opportunistic pathogen with innate resistance to many antibiotics. In places that are economically backward, these problems get compounded by the inability of patients to afford newer expensive drugs. Topically applied dilute acetic acid, which is cheap and easily available, has been found to be effective in such chronic wounds. They pose a major challenge that is cumbersome in terms of wound healing and also add to the cost in terms of quality of life to the patient and is a financial burden for the hospitals. Three main factors have been found to be the causative factors for the development of a chronic wound: firstly, bacterial colonisation or commonly called bioburden; secondly, reperfusion injury; and thirdly, cellular and systemic factors. Most of the wounds if not all of them are contaminated with pathogenic microorganisms, but this itself does not affect the healing of wounds. When the contamination increases to a point of critical colonisation or infection, then the infection or the bioburden in the wound becomes a major contributing factor that impedes wound healing. Chronic wounds do not progress to the proliferative phase of wound healing and undergo a detention in the inflammatory phase of healing because of which there is a continuous influx of neutrophils into the wound area, with the release of free radicals, cytolytic enzymes and inflammatory mediators that cause damage to the invading pathogens as well as to the host tissue. Poor blood supply results in hypoxic conditions in tissues, which can lead to cell death and tissue necrosis. This provides good growing conditions for pathogenic microorganisms leading to the establishment and colonisation of bacteria in the host tissue.

ELIGIBILITY:
Inclusion Criteria:

* Chronic diabetic wounds
* All gender
* age 40-65 years

Exclusion Criteria:

* Chronic wounds due to trauma, neoplasm, burn
* peripheral vascular disease
* Osteomyelitis grade 3 and above.

Data collection:

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Early epithelialization and granulation | at 48 hours, 72 hours and 07 days
  After selection of the patients adequate antibiotics were given as per standard hospital protocol. Patients were assessed for application of 1% acetic acid dressing after every 12 hours for early epithelialization and granulation which will be diagnosed clinically by examining the wound respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Pak Emirates military hospital, Rawalpindi, Punjab Province, Pakistan